CLINICAL TRIAL: NCT06910735
Title: Effect of Financial Incentives on Weight Loss in Patients With Failed Bariatric Surgery: A Multicenter Randomized Open-Label Trial
Brief Title: Financial Incentives and Weight Loss in Failed Bariatric Surgery
Acronym: BARIACADO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: APHP220835; PREPS-21-0030 (Other Grant/Funding Number: French Ministry of Health); 2023-A01309-36 (Other: Agence nationale de sécurité du médicament et des produits de santé); 23.02108.000240 (Other: Commission Nationale des Recherche Impliquant la Personne Humaine)
Record Dates: First submitted 2025-03-28; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Obesity; Obesity Recidivism
Keywords: Bariatric surgery; Financial incentive
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Other)
  Interventions: Other: Control
- Threshold financial incentive (Experimental)
  Interventions: Behavioral: Threshold financial incentive
- Proportional financial incentive (Experimental)
  Interventions: Behavioral: Proportional financial incentive

INTERVENTIONS:
Other: Control — Participants will receive the standard care that includes setting a weight-loss target based on the weight achieved at 12 months post-bariatric surgery following the standard multidisciplinary follow-up at the inclusion center
  Arms: Control
Behavioral: Threshold financial incentive — Participants will receive the standard care with an additional financial incentive of 300 € if they successfully achieve the weight loss target corresponding to their weight at 12 months after bariatric surgery. This financial incentive will be awarded 12 months after their inclusion in the study.
  Arms: Threshold financial incentive
Behavioral: Proportional financial incentive — Participants will receive the standard care with an additional financial incentive, which will be determined based on the proportion of their actual weight loss in relation to the predefined weight loss target corresponding to their weight at 12 months after bariatric surgery. The financial incentive can be up to 300 € if the weight loss target is achieved 12 months after their inclusion in the study.
  Arms: Proportional financial incentive

SUMMARY:
This national, prospective, multicenter, and randomized study seeks to evaluate the effect of financial incentives on weight loss in individuals who experience weight regain following bariatric surgery. The study also aims to conduct a cost-utility analysis to measure the effectiveness of the intervention and assess the potential budgetary implications if it were to be implemented on a wider scale.

DETAILED DESCRIPTION:
Our intervention is based on the principle of "contingency management" whereby financial rewards are contingent upon meeting specific weight loss targets. To assess the effectiveness of this approach, patients who have experienced weight regain after bariatric surgery will be randomly assigned to one of three groups. Group 1 will receive the standard care that includes setting a weight-loss target based on the weight achieved at 12 months post-bariatric surgery following the standard multidisciplinary follow-up at the inclusion center. Group 2 will receive the same treatment as the control group (Group 1), but with an additional financial incentive if the weight loss target (corresponding to the weight they reached 12 months after bariatric surgery) is achieved 12 months after inclusion. Group 3 will receive the same treatment as the control group (Group 1), but the financial incentive will be proportional to the actual weight loss achieved relative to the weight loss target (corresponding to the weight they reached 12 months after bariatric surgery).

The study will include a standard post-bariatric surgery follow-up visits scheduled at 6, 12, 18, and 24 months, as per routine practice. At the 12-month visit, participants will be eligible to receive a financial incentive based on their arm assignment and the extent of weight loss achieved. After the 12-month visit, participants will not receive any additional financial incentives until the 24-month visit.

ELIGIBILITY:
Inclusion Criteria:

* Male or female over 18 years of age
* Patients with a history of adjustable gastric banding, sleeve gastrectomy, gastric bypass or SADI-sleeve surgery
* Patient with a post-operative delay of more than 2 years
* Patient who has gained ≥10% of the maximum weight lost
* Patient still obese (body mass index ≥ 30 kg/m²) after surgery

Exclusion Criteria:

* Pregnant women
* Women of childbearing potential planning a pregnancy during the first year of the study
* Persons under legal protection (safeguard of justice, guardianship, curatorship, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2028-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in body weight | 12 months

SECONDARY OUTCOMES:
Change from Baseline in body weight | 24 months
Change from Baseline in blood pressure | 6, 12, 18, 24 months
Change from Baseline in Fasting Plasma Glucose | 6, 12, 18, 24 months
Change from Baseline in Glycated hemoglobin | 6, 12, 18, 24 months
Change from Baseline in Total Cholesterol | 6, 12, 18, 24 months
Change from Baseline in High-density Lipoproteins | 6, 12, 18, 24 months
Change from Baseline in Low-density Lipoproteins | 6, 12, 18, 24 months
Change from Baseline in Triglycerides | 6, 12, 18, 24 months
Change from Baseline in AST levels | 6, 12, 18, 24 months
Change from Baseline in ALT levels | 6, 12, 18, 24 months
Change from Baseline in the adherence to multivitamins intake | 6, 12, 18, 24 months
Change from Baseline in quality of life as measured by the Moorehead-Ardelt questionnaire | 6, 12, 18, 24 months
Change from Baseline in quality of life as measured by the EQ-5D-5L questionnaire | 6, 12, 18, 24 months
Rate of participants who achieve the predefined weight loss target | 12, 24 months
Difference in incremental cost-effectiveness ratio | 12, 24 months
Difference in the costs generated to the healthcare system | 12, 24 months
Difference in the costs avoided to the healthcare system | 12, 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien Czernichow, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (12):
- France (12):
  - AP-HP - hôpital Avicenne, Bobigny
  - AP-HP - hôpital Louis-Mourier, Colombes
  - Centre hospitalier intercommunal de Créteil, Créteil
  - AP-HM - hôpital de la Conception, Marseille
  - CHU de Nantes - hôpital Laënnec, Nantes
  - CHR d'Orléans - hôpital La Source, Orléans
  - AP-HP - hôpital de la Pitié-Salpêtrière, Paris
  - AP-HP - hôpital européen Georges-Pompidou, Paris
  - AP-HP - hôpital Bichat - Claude-Bernard, Paris
  - CHU de Poitiers, Poitiers
  - CHU de Reims - hôpital Robert-Debré, Reims
  - CHU de Nancy - hôpital Brabois, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in publication could be shared. IPD detailed in the protocol of a planned metaanalysis could be shared.
Supporting Information: Study Protocol, ICF
Time Frame: Two years after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI based on a scientific project and scientific involvement of the PI team. Collaboration will be fostered.
  Teams wishing obtain IPD must meet the sponsor and IP team to present scientifics (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory contractualization.
  Processing of shared data must comply with European General Data Protection Regulation (GDPR).